CLINICAL TRIAL: NCT04207489
Title: Prospective Registry Study of Endoscopic Submucosal Injection of Indocyanine Green Before Laparoscopic Radical Resection for Colorectal Cancer
Brief Title: Endoscopic Submucosal Injection of Indocyanine Green Before Laparoscopic Radical Resection for Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Dong Yang, Assisted Investigator, Jilin University
Other Study IDs: 130003
Record Dates: First submitted 2019-12-17; First posted 2019-12-23 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer; Indocyanine Green
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endoscopic submucosal injection of indocyanine green
  Interventions: Procedure: endoscopic submucosal injection of indocyanine green before laparoscopic radical operation of colorectal cancer

INTERVENTIONS:
Procedure: endoscopic submucosal injection of indocyanine green before laparoscopic radical operation of colorectal cancer — Indocyanine green was injected under endoscope within 24 hours before operation. Four points were evenlyinjected in four quadrants at the edge of the tumor. The patients with obstruction were injected at two points on the anal side of the tumor. The diluted concentration of indocyanine green was 0.625mg/ml or 1.25mg/ml. The injection method was direct submucosal injection and sandwich method. According to the imaging effect, it can be divided into local imaging and lymphatic drainage imaging. Tumor body: 0, no imaging; 1, full imaging; 2, diffuse imaging, overflow, interference with other areas of observation. Lymph drainage area imaging 0, no imaging; 1, full imaging; 2, diffuse imaging, overflow, interference with other areas of observation.

SUMMARY:
Prospective registry study of endoscopic submucosal injection of indocyanine green before laparoscopic radical resection for colorectal cancer

DETAILED DESCRIPTION:
To observe the imaging result of endoscopic submucosal injection of indocyanine green before laparoscopic radical resection for colorectal cancer, and analyze the relevant factors, so as to guide the submucosal injection of preoperative indocyanine green better.

This study is prospective and observational. In order to analyze the related factors that affect the imaging effect, we enrolled patients who were to undergo indocyanine green fluorescence imaging for laparoscopic radical resection for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were to undergo indocyanine green fluorescence imaging for laparoscopic radical operation of colorectal cancer.

Exclusion Criteria:

* have simultaneously other cancer

  * have severe systemic inflammatory disease ,serious illness such as diabetes, chronic lung diseases
  * have gastrointestinal surgery
  * Indocyanine green or iodine allergy
  * the period is too late or the tumor is too large to carry on a laparoscopic surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were to undergo indocyanine green fluorescence imaging for laparoscopicradical operation of colorectal cancer.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-12-25 (Estimated); Study Completion 2021-04-28 (Estimated)

PRIMARY OUTCOMES:
The imaging effect of indocyanine green | During the operation
  The imaging effect was evaluated by indocyanine green fluorescence imaging system during the operation. According to the imaging effect, it can be divided into local imaging and lymphatic drainage imaging. Tumor body: 0, no imaging; 1, full imaging; 2, diffuse imaging, overflow, interference with other areas of observation. Lymph drainage area imaging 0, no imaging; 1, full imaging; 2, diffuse imaging, overflow, interference with other areas of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Yang, Master, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No